CLINICAL TRIAL: NCT00807573
Title: A Phase II Trial of Paclitaxel, Bevacizumab and Pemetrexed in Patients With Untreated, Advanced Non-Small Cell Lung Cancer Using Web-Based Data Collection, Patient Self-Reporting of Adverse Effects and Automated Response Assessment
Brief Title: Paclitaxel, Bevacizumab and Pemetrexed in Patients With Untreated, Advanced Non-Small Cell Lung Cancer Using Web-Based Data Collection, Patient Self-Reporting of Adverse Effects and Automated Response Assessment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-109
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: BEVACIZUMAB (AVASTIN); PEMETREXED (ALTIMA); TAXOL (PACLITAXEL); 08-109
MeSH Terms: conditions — Lung Neoplasms | interventions — Paclitaxel; Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel, Bevacizumab & Pemetrexed (Experimental): During each 28-day cycle, paclitaxel, pemetrexed and bevacizumab will be given intravenously on days 1 and 15. Paclitaxel will be administered at 90mg/m^2 over 60 minutes on days 1 and 15. Pemetrexed 500mg/m^2 will be administered over 10 minutes on days 1 and 15. Bevacizumab will be given at 10mg/kg over 20 minutes on days 1 and 15
  Interventions: Drug: Paclitaxel; Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Day 1: Paclitaxel (90 mg/m^2 over 60 minutes) Day 15: Paclitaxel (90 mg/m^2 over 60 minutes)
Drug: Pemetrexed — Day 1: Pemetrexed (500 mg/m^2 over 10 minutes) Day 15 Pemetrexed (500 mg/m2 over 10 minutes)
Drug: Bevacizumab — Day 1:Bevacizumab (10 mg/kg over 20 minutes) Day 15: Bevacizumab (10 mg/kg over 20 minutes)

SUMMARY:
The purpose of this study is to determine the percentage of patients with non-small cell lung cancer that will experience a shrinkage of their tumors following treatment with three medications given together: paclitaxel, pemetrexed (Alimta®), and bevacizumab (Avastin®). Each of these medications has been approved by the FDA for patients that have not received any treatment for their lung cancer. This study is designed to study the effects of all three drugs given at the same time.

Each of these medications has been studied in lung cancer and is commercially available. Paclitaxel and pemetrexed are traditional chemotherapy drugs. Bevacizumab is a monoclonal antibody, which means that it attaches to a specific target. Bevacizumab attaches to a protein in the blood stream called Vascular Endothelial GrowthFactor (VEGF). VEGF helps tumors grow new blood vessels to feed themselves, and bevacizumab is thought to help block this new growth of blood vessels and starve the tumors of the nutrients they need.

DETAILED DESCRIPTION:
In this clinical trial, we also will be studying other things. We want to learn more about how to manage side effects patients may develop during chemotherapy. Cancer patients may develop side effects during treatment, such as nausea, pain, fatigue, diarrhea, constipation, or shortness of breath. These symptoms may be due to the cancer itself, or due to treatments like chemotherapy drugs or radiation therapy. Doctors and nurses often ask patients about their symptoms, because an important part of cancer treatment is to make patients feel as well as possible. If patients do not feel well, we may need to change the way we are treating them or prescribe therapies that will decrease their symptoms. The best way to find out how the patient is feeling is to ask them directly.

We are interested in developing new ways to ask patients about how they are feeling, using the Internet. A special new website called STAR ("Symptom Tracking and Reporting for Patients") has been developed to help patients record this information, so that their doctors and nurses can review it during clinic appointments. This study is designed to help us see if STAR is a helpful way for us to keep track of information about patients' symptoms and quality of life.

As part of this study, a computerized (automated) technique of determining the size of the patients tumor(s) before and after treatment will be used. This has been tested in the past and found to be more accurate. The automated technique of determining tumor size will be used with the routine CT scans that the patient will have as part of the study. This automated method of measuring the tumor(s) will allow us to know sooner whether this drug treatment is causing the disease to shrink.

The information from STAR and the automated tumor measurements are going to be placed on a very secure Internet site. This will provide the doctor with all of the information needed to determine if this drug combination is working for the patient and whether to continue this study.

Also, if there is a tumor sample from a biopsy done in the past, it will be analyzed for a protein that may be present in the lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Non-Small Cell Lung Cancer at MSKCC
* Clinical stage IIIB or IV.
* Measurable disease as per RECIST
* Greater than 6 months since receiving neo-adjuvant or adjuvant chemotherapy for Non-Small Cell Lung Cancer.
* Age ≥ 18 years.
* Karnofsky performance status of ≥ to 70.
* Marrow and organ function as follows:
* WBC ≥ to 4000/mm3
* Platelets ≥ to 160,000
* Bilirubin ≤ to 1.2mg/dL
* Creatinine clearance ≥ to 40mL/min
* AST and/or /ALT ≤ 37 Units/L (if one of these elevated, must be ≤ 2.5 ULN)
* Systolic blood pressure ≤ to 150mmHg or diastolic blood pressure ≤ to 100 mmHg).
* The subject is able to read and comprehend English text from a computer screen.
* Women of childbearing potential and sexually active men enrolled in the study must agree to practice effective contraception.

Exclusion Criteria:

* Squamous cell carcinoma.
* Prior treatment with paclitaxel, pemetrexed or bevacizumab for NSCLC.
* Prior systemic anticancer therapy for advanced NSCLC.
* Symptomatic brain metastases with evidence of hemorrhage.
* Radiation therapy to greater than 25% of the bone marrow within 30 days of starting treatment.
* Peripheral neuropathy greater than grade 1.
* Malignancies within the past 5 years other than non-melanoma skin cancer.
* Patients with other serious medical illnesses including, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of hemoptysis.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess.
* History of myocardial infarction or stroke within 6 months prior to enrollment.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pietanza, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- [Derived] Basch E, Wood WA, Schrag D, Sima CS, Shaw M, Rogak LJ, Kris MG, Shouery M, Bennett A, Atkinson T, Pietanza MC. Feasibility and clinical impact of sharing patient-reported symptom toxicities and performance status with clinical investigators during a phase 2 cancer treatment trial. Clin Trials. 2016 Jun;13(3):331-7. doi: 10.1177/1740774515615540. Epub 2015 Nov 4. PMID 26542025
- [Derived] Pietanza MC, Basch EM, Lash A, Schwartz LH, Ginsberg MS, Zhao B, Shouery M, Shaw M, Rogak LJ, Wilson M, Gabow A, Latif M, Lin KH, Wu Q, Kass SL, Miller CP, Tyson L, Sumner DK, Berkowitz-Hergianto A, Sima CS, Kris MG. Harnessing technology to improve clinical trials: study of real-time informatics to collect data, toxicities, image response assessments, and patient-reported outcomes in a phase II clinical trial. J Clin Oncol. 2013 Jun 1;31(16):2004-9. doi: 10.1200/JCO.2012.45.8117. Epub 2013 Apr 29. PMID 23630218
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel, Bevacizumab & Pemetrexed: Paclitaxel, Bevacizumab and Pemetrexed in Untreated, Advanced Non-Small Cell Lung Cancer. During each 28-day cycle, paclitaxel, pemetrexed and bevacizumab will be given intravenously on days 1 and 15. Paclitaxel will be administered at 90mg/m^2 over 60 minutes on days 1 and 15. Pemetrexed 500mg/m^2 will be administered over 10 minutes on days 1 and 15. Bevacizumab will be given at 10mg/kg over 20 minutes on days 1 and 15, and 19.
Period: Overall Study
Arm/Group | Paclitaxel, Bevacizumab & Pemetrexed
Started | 44
Completed | 42
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel, Bevacizumab & Pemetrexed: Paclitaxel, Bevacizumab and Pemetrexed in Untreated, Advanced NSCLC. During each 28-day cycle, paclitaxel, pemetrexed and bevacizumab will be given intravenously on days 1 and 15. Paclitaxel will be administered at 90mg/m2 over 60 minutes on days 1 and 15. Pemetrexed 500mg/m2 will be administered over 10 minutes on days 1 and 15. Bevacizumab will be given at 10mg/kg over 20 minutes on days 1, 15 and 19.
Arm/Group | Paclitaxel, Bevacizumab & Pemetrexed
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (CR + PR by RECIST) Paclitaxel, Pemetrexed, and Bevacizumab in Patients With Advanced Non-Small Lung Cancer Who Have Received no Prior Treatment for Metastatic Disease.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Paclitaxel, Bevacizumab & Pemetrexed
Number analyzed (Participants) | 42
participants
  Partial Response | 27
  Stable Disease | 15

ADVERSE EVENTS:
Arm/Group | Paclitaxel, Bevacizumab & Pemetrexed
Serious Adverse Events (participants affected / at risk) | 20/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, Bevacizumab & Pemetrexed (N=44)
Death not assoc w CTCAE term- Death NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema: limb (General disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Hemoglobin (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 2 (3)
Infection, other (Infections and infestations) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy: cranial - CN II Vision (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Perforation, GI- Small Bowel NOS (Gastrointestinal disorders) | 1 (1)
Pneumonitis/pulm infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Vessel injury-artery- Other NOS (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel, Bevacizumab & Pemetrexed (N=44)
ALT, SGPT (Investigations) | 21 (116)
AST, SGOT (Investigations) | 11 (32)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13 (37)
Anorexia (Metabolism and nutrition disorders) | 21 (70)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (35)
Creatinine (Investigations) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 22 (84)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 30 (213)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 35 (176)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 10 (49)
Hemoglobin (Investigations) | 18 (123)
INR (Investigations) | 2 (8)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 21 (87)
Lymphopenia (Blood and lymphatic system disorders) | 19 (162)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 10 (26)
Nausea (Gastrointestinal disorders) | 11 (35)
Neuropathy: sensory (Nervous system disorders) | 9 (21)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 18 (45)
PTT (Investigations) | 2 (2)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 21 (66)
Pain - Pain NOS (General disorders) | 28 (143)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 8 (13)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (9)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 4 (5)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (7)
Voice changes/dysarthria (Nervous system disorders) | 8 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes